CLINICAL TRIAL: NCT05965778
Title: Comparison of the Performance and Safety of T2769 Versus Vismed® Multi in the Treatment of Moderate to Severe Dry Eye Syndrome
Brief Title: Performance and Safety of T2769 in DED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT2769-002
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Change from baseline in the study eye at Day 36 in Global Ocular staining (decrease of oxford score = better outcome)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T2769 (Experimental): 1 drop in each eye, 3 to 6 times daily
  Interventions: Device: T2769
- Vismed® Multi (Active Comparator): 1 drop in each eye, 3 to 6 times daily
  Interventions: Device: Vismed® Multi

INTERVENTIONS:
Device: T2769 — T2769: sodium hyaluronate, Trehalose, Naaga in a 12.5 mL ABAK® multi-dose bottle.
  Arms: T2769
Device: Vismed® Multi — Hyaluronic acid
  Arms: Vismed® Multi

SUMMARY:
To demonstrate the non-inferiority of T2769 compared to Vismed® Multi in terms of total ocular surface staining (Oxford score) after 35 days of treatment.

To evaluate the performance and safety of T2769 versus Vismed® Multi.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated (obtained prior to initiating any procedures).
* Patient aged ≥18 years old.
* Known dry eye syndrome requiring artificial tears for at least the last 3 months prior to screening visit.
* Surface Disease Index (OSDI) Score ≥ 23.
* Ocular discomfort evaluated by VAS ≥ 40 mm.

Exclusion Criteria:

* Far best-corrected visual acuity (BCVA) ≥+0.7 LogMar (e.g., ≤0.2 in decimal value or ≤20/100 Snellen equivalent or ≤50 (ETDRS) letters Early Treatment Diabetic Retinopathy Study).
* Severe blepharitis according to the judgment of the investigator
* Dry eye associated with at least one of the following diseases/symptoms: ocular rosacea, Pterygium, Eyelid malposition, Corneal dystrophy, Ocular neoplasia, Filamentous keratitis, Corneal neovascularisation, Orbital radiotherapy, Cataract, Retinal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric CHIAMBARETTA, Prof., Principal Investigator — Individual Practice for Specialized Ophthalmology Care
Locations (1):
- Gabriel-Montpied University Hospital, Clermont-Ferrand, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T2769 | Vismed® Multi
Started | 125 | 126
Completed | 113 | 111
Not Completed | 12 | 15
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — divers reasons(patient or doctor not available for visit...), | 9 | 7

BASELINE CHARACTERISTICS:
Population: ITT set
Groups:
- Total: Total of all reporting groups
Arm/Group | T2769 | Vismed® Multi | Total
Number analyzed (Participants) | 125 | 126 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 76 | 150
  >=65 years | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (15.04) | 60.1 (13.64) | 59.4 (14.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 104 | 204
  Male | 25 | 22 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 3 | 0 | 3
  Austria | 15 | 15 | 30
  Spain | 43 | 46 | 89
  Greece | 14 | 13 | 27
  Hungary | 6 | 5 | 11
  Israel | 16 | 16 | 32
  Italy | 11 | 17 | 28
  Slovakia | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Surface Ocular Staining With Fluorescein (With Oxford Scale - Ranges : Minimum 0- Maximum 15)
Description: Change from baseline (Day 1) in the worse eye at Day 36 in Global Ocular staining (decrease of oxford score = better outcome)
Time Frame: Oxford 0-15 grading scheme: is assessed at Day 1 and Day 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T2769 | Vismed® Multi
Number analyzed (Participants) | 123 | 121
score on a scale | -2.3 (1.99) | -2.1 (2.08)

ADVERSE EVENTS:
Time Frame: 7 weeks from D-10 to D36 (+3 days)
Arm/Group | T2769 | Vismed® Multi
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/125 | 2/126
Other Adverse Events (participants affected / at risk) | 0/125 | 0/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T2769 (N=125) | Vismed® Multi (N=126)
Limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Hand phalanx fracture
haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) — Macroscopic haematuria

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT05965778/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT05965778/SAP_001.pdf